CLINICAL TRIAL: NCT00948636
Title: A Multicenter Study of Hematopoietic Stem Cell Donor Safety and Quality of Life
Brief Title: Stem Cell Related Donor Safety Study
Acronym: RDSafe
Status: Completed | Type: Observational
Sponsor: Center for International Blood and Marrow Transplant Research (Network)
Collaborators: National Institutes of Health (NIH) (NIH); University of Utah (Other); University of Pittsburgh (Other)
Responsible Party: Sponsor
Other Study IDs: 06-DON
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Last update posted 2017-06-14 (Actual); Status verified 2016-07

CONDITIONS: Related Hematopoietic Stem Cell Donors

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Related Donors: Related Hematopoietic Stem Cell Donors

SUMMARY:
The study tests the hypothesis that related hematopoietic stem cell donors are at a higher risk for acute medical and psychological toxicity associated with the donation process compared to adult unrelated hematopoietic stem cell donors.

The study will also assess the hypothesis that young (<18 years) and older (>60 years) related donors are at increased risk for toxicity associated with donation compared to younger adult donors by describing the adverse events reported in these populations.

An ancillary study of the psychological impact of donation on health-related quality of life (HRQoL) will enroll related donors and compare them to an age-matched normative cohort.

ELIGIBILITY:
Inclusion Criteria:

* Donors of any age providing either a first or second BM or PBSC donation
* Meet donation criteria per institution policies and procedures
* Willing to receive phone follow-up at 1, 6, and 12 months
* Signed informed consent for study participation

For the HRQoL ancillary study, inclusion criteria:

* Related donors age greater than or equal to 5, eligible and consented to the primary trial by the above listed inclusion criteria
* Donors competent to answer psychological assessment questions by themselves, or if a child, should be able to respond to psychological assessment questions and have an appropriate proxy also able to complete the HRQoL proxy interview
* English speaking
* Access to a telephone
* Willing to participate in pre-donation, 1 month and 1 year follow-up interviews
* Signed informed consent for study participation in ancillary study

Exclusion Criteria:

* Per institutional guidelines
* Donors providing unstimulated peripheral blood stem cells or lymphocytes

For the HRQoL ancillary study, exclusion criteria:

* Children less than or equal to 4 years of age

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: participating institutions (transplant centers)
Sampling Method: Non-Probability Sample
Enrollment: 1812 (Actual)
Dates: Start 2010-01; Primary Completion 2015-08 (Actual); Study Completion 2016-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael A Pulsipher, M.D., Principal Investigator — Children's Hospital Los Angeles
Locations (52):
- United States (52):
  - Banner Good Samaritan Medical Center, Phoenix, Arizona
  - University of California, San Diego, San Diego, California
  - University of California, San Francisco, San Francisco, California
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Florida Center for Cellular Therapy, Orlando, Florida
  - All Children's Hospital, St. Petersburg, Florida
  - H. Lee Moffitt Cancer Center, Tampa, Florida
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Winship Cancer Institute, Atlanta, Georgia
  - Children's Memorial Medical Center, Chicago, Illinois
  - University of Chicago, Chicago, Illinois
  - Indiana Blood and Marrow Transplantation, LLC, Beech Grove, Indiana
  - Riley Hospital for Children, Indianapolis, Indiana
  - University of Iowa Hospitals, Iowa City, Iowa
  - University of Kansas Medical Center, Westwood, Kansas
  - Kosair Children's Hospital, Louisville, Kentucky
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMass Memorial Medical Center, Worcester, Massachusetts
  - University of Michigan Medical Center, Ann Arbor, Michigan
  - Barbara Ann Karmanos Cancer Center, Detroit, Michigan
  - Helen DeVos Children's Hospital - Spectrum Health, Grand Rapids, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, Rochester, Minnesota
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University, St Louis, Missouri
  - John Theurer Cancer Center - Hackensack University Medcial Center, Hackensack, New Jersey
  - Roswell Park Cancer Institute, Buffalo, New York
  - North Shore University Hospital, Lake Success, New York
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Mt. Sinai Medical Center, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - University of Rochester Medical Center, Rochester, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Duke University Medical Center, Durham, North Carolina
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina
  - Jewish Hospital, Cincinnati, Ohio
  - University Hospitals of Cleveland/Case Western, Cleveland, Ohio
  - Cleveland Clinic, Cleveland, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oregon Health and Science University, Portland, Oregon
  - Penn State Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - The Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - University of Texas Southwestern Medical Center, Dallas, Texas
  - Texas Institute of Medicine and Surgery, San Antonio, Texas
  - University of Utah, Primary Children's Medical Center, Salt Lake City, Utah
  - University of Utah, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Fred Hutchinson Cancer Research Center, Seattle, Washington
  - University of Wisconsin, Madison, Wisconsin
  - Medical College of Wisconsin, Milwaukee, Wisconsin